CLINICAL TRIAL: NCT05588154
Title: Collection of Blood, Bone Marrow, Skin, Saliva, and Stool Samples From Healthy Volunteers Used for Comparative Analysis of Myeloid Malignancies
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000975; 000975-C
Record Dates: First submitted 2022-10-19; First posted 2022-10-20 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12-04

CONDITIONS: Myelodysplastic Syndromes
Keywords: Hematopoietic Stem Cell Malignancies; Acute Myeloid Leukemia; DNA methyltransferase inhibitors; Treatment-Related Complications; Cytotoxic Therapy; Natural History
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Healthy volunteers who will donate blood, and/or bone marrow and may donate other samples
- Cohort 2: Healthy volunteers who will donate stool samples only

SUMMARY:
Background:

Myelodysplastic syndromes (MDS) are disorders of blood stem cells that can develop into blood cancers. Treatment options are limited. To find better treatments, researchers need to better understand how MDS develops. To do that, they must be able to compare biospecimens from people with the disease to those of healthy people.

Objective:

This study will create a database of biospecimens collected from healthy volunteers.

Eligibility:

Healthy people aged 18 and older.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests.

Up to 5 types of samples will be collected on 1 or more days within 1 month of screening:

Blood: Blood will be drawn by inserting a needle into a vein.

Saliva: Participants will scrape the insides of their cheeks with a brush.

Stool: Participants will be given a container to collect stool at home. They will use a prepaid envelope to mail in the sample.

Bone marrow: A sample of the soft tissue inside the bones will be drawn out. The area to be biopsied, usually the lower back, will be numbed. A needle will be inserted through a small cut to remove the sample. Participants' pain will be monitored; additional numbing medicine may be used.

Skin: A piece of skin about 1/6 of an inch across will be cut away. Stitches may be used to close the wound. Participants will return to the clinic to have the stitches removed.

Participants do not have to provide all of the samples listed. They will give each sample only once.

DETAILED DESCRIPTION:
Background:

* Myelodysplastic syndromes (MDS) are heterogeneous stem cell disorders characterized by ineffective hematopoiesis resulting in cellular dysplasia, peripheral cytopenias, and increased risk for transformation to acute myeloid leukemia (AML).
* There are limited treatment options, all of which have unimpressive response rates and limited response durations, with the only potential cure being hematopoietic stem cell transplant (HSCT). Unfortunately, as a disease of the elderly (average age of diagnosis >65 years), most participants are not eligible for HSCT due to advanced age and other comorbidities.
* It is critical we further elucidate the processes that lead to disease manifestation to develop novel therapeutic strategies and alter the natural history of the disease.
* In order to understand the biology of the disease, it is critical to have control biospecimens from healthy individuals to delineate the mechanisms driving disease pathogenesis.

Objective:

-To create a database of analyzed biospecimens collected from healthy volunteers.

Eligibility:

* Age >= 18 years old
* Healthy volunteers as confirmed by clinical evaluation

Design:

* This is a trial to analyze samples from healthy volunteers collected at NIH Clinical Center.

  --Participants = will be asked to provide blood, and/or bone marrow, and other samples (skin biopsy samples, saliva, stool samples).
* The total protocol accrual goal is 1,000 participants. Enrollment is expected to take place over approximately 20-50 years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age >= 18 years old
* Healthy volunteers; the following confirmed by the Principal Investigator or designees based on recent (within 3 months before study intervention(s))
* medical history
* physical exam
* complete blood count (CBC) within the normal reference range per the reporting clinical laboratory, established published literature and reports, or as deemed acceptable by the medical team based on the age and condition of the volunteer consistent with established clinical standards.
* The ability of the participant to understand and the willingness to sign a written consent document.

EXCLUSION CRITERIA:

- Active illnesses, immunodeficiency, history of opportunistic infection, autoimmune disease, history of or active malignancy, prior organ, bone marrow, or peripheral blood stem cell transplant or antibiotic treatment within 3 months before study intervention(s).

Note: participants with non-melanoma skin cancer or carcinoma in situ of the cervix or breast are eligible.

* Current immunosuppressive medication.
* Any one of the following symptoms as declared by the participant at least one day per week within 3 months before study intervention(s) (Rome IV criteria [36])
* Diarrhea characterized as frequent (>2) loose stools
* Constipation defined as < 3 spontaneous bowel movements per week
* Bloating and/or distention
* Abdominal pain.
* Participants with a history of the human immunodeficiency virus (HIV), hepatitis C (HCV), or hepatitis B (HBV) as confirmed by a seropositive blood test.
* Pregnancy confirmed with beta-Human Chorionic Gonadotropin (Beta-HCG) serum or urine pregnancy test performed in women of childbearing potential at screening.
* Breastfeeding participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are healthy volunteers, selected from the general population. Employees may also volunteer per the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2052-12-01 (Estimated); Study Completion 2052-12-01 (Estimated)

PRIMARY OUTCOMES:
create a database of analyzed biospecimens | ongoing
  Collection of biospecimens from healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy L McGraw, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All large scale genomic sequencing data will be shared with subscribers to dbGaP.@@@@@@All collected IPD will be shared via request to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.@@@@@@Non genomic clinical data will be shared 10 years after the primary objective has been attained
Access Criteria: Genomic data are made available via dbGaP through requests to the data custodians.@@@@@@The principal investigator will review IPD requests.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000975-C.html